CLINICAL TRIAL: NCT01743196
Title: Pilot Study of Folate Pharmacokinetics in Normal Weight and Obese Women of Child-bearing Age
Brief Title: Folate Metabolism in Normal Weight and Obese Women of Child-bearing Age
Status: Completed | Type: Observational
Sponsor: University of Georgia (Other)
Responsible Party: Principal Investigator, Lynn B. Bailey, PhD, Department Head and Professor, University of Georgia
Other Study IDs: UGAFOLATEPILOT
Record Dates: First submitted 2012-12-04; First posted 2012-12-06 (Estimated); Last update posted 2015-10-21 (Estimated); Status verified 2015-10

CONDITIONS: Obesity; Neural Tube Defects
Keywords: Folic acid; Folate; Pharmacokinetics; Women of Child Bearing Age
MeSH Terms: conditions — Obesity; Neural Tube Defects

STUDY DESIGN:
Biospecimen Retention: Samples With DNA — Buffy Coat Serum samples Plasma samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Normal weight: Women with BMI 18.5 to 24.9 kg/m2
- Obese: Women with BMI > 30 kg/m2

SUMMARY:
The purpose of this study is to determine if there is a difference in the short term response in serum folate after a single dose of folic acid in normal weight and obese women of childbearing age.

DETAILED DESCRIPTION:
Current recommendations established in 1998, specify that all women capable of becoming pregnant consume 400 micrograms of folate daily from supplements, fortified foods, or both, in addition to consuming food folate from a varied diet. Despite this recommendation, obese women have a lower folate status than women of normal weight which suggests that obesity may have a negative impact on folate metabolism. Therefore, the objective of this study is to determine if there are differences in the metabolic response to a single dose of folate between normal weight and obese women of child bearing age. The two groups of women will be given the currently recommended amount of folic acid, 400 micrograms, and blood samples will be taken before the vitamin is given and at various points afterwards to determine serum folate response to the folate dose. Results of this research should help determine if folate requirements are higher for obese than for non-obese women. The long-term goal of this and follow-up studies is to generate data that will contribute to the evidence base used by scientific advisory panels to determine whether dietary folate intake recommendations should be based on body weight.

ELIGIBILITY:
Inclusion Criteria:

* Female 18-35 yr
* Caucasian
* Body mass index 18.5 - 24.9 or > 30 kg/m2

Exclusion Criteria:

* Currently pregnant, pregnancy within the past 12 months
* Greater than 2 previous pregnancies
* Use of prescription drugs other than oral contraceptives
* Chronic disease (diabetes, hypertension, epilepsy, cancer, kidney disease, cardiovascular disease)
* Acute illness (e.g. pneumonia, urinary tract infection, mononucleosis)
* Use of antibiotics in past 30 days
* Current smoker
* Use of dietary supplements including multivitamins in the past 30 days
* Significant weight change in past 12 months
* Typical alcohol consumption of 2 or more drinks per day
* Consumption of any alcohol in the week preceding testing

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Community sample from Athens, GA and surrounding area
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2012-05; Primary Completion 2012-08 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Area under the serum concentration versus time curve (AUC) for folic acid | 0, 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 4.0, 5.0, 6.0, 7.0, 8.0, 9.0 10.0 hours post-dose
  Change from baseline in serum folate response at the indicated time points following oral intake of a 400 ug dose of folic acid will be calculated by subtracting the baseline concentrations from the folate value at each subsequent time point. Individual response-time curves will be generated and area-under-the-curve (AUC) calculated using the trapezoidal rule.

SECONDARY OUTCOMES:
Peak Serum Concentration (Cmax) of Folate | up to 10 hours
  Maximum folate concentration in response to an oral dose of 400 ug folic acid. Values are derived from the individual response curves.
Time to peak concentration (tmax) of folate | up to 10 hours
  Time to peak serum concentration of folate following the oral administration of a 400 ug dose of folic acid. Values are derived from the individual response curves.

CONTACTS AND LOCATIONS:
Overall Officials: Lynn B Bailey, PhD, Principal Investigator — University of Georgia
Locations (1):
- University of Georgia, Athens, Georgia, United States

REFERENCES:
- [Result] da Silva VR, Hausman DB, Kauwell GP, Sokolow A, Tackett RL, Rathbun SL, Bailey LB. Obesity affects short-term folate pharmacokinetics in women of childbearing age. Int J Obes (Lond). 2013 Dec;37(12):1608-10. doi: 10.1038/ijo.2013.41. Epub 2013 Apr 9. PMID 23567925